CLINICAL TRIAL: NCT01060995
Title: SmartConsent: A Computerized Informed Consent for Patients
Acronym: SmartConsent
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Center for Clinical and Translational Sciences (CCTS) Clinical Research Unit at The University of Texas Health Science Center at Houston (Other)
Responsible Party: Principal Investigator, John Valenza, Dean and Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-DB-07-0593
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: Informed Consent; Oral Health; Patient Decision-making

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SmartConsent: Subjects receiving SmartConsent informed consent
- Standard consent: Subjects receiving standard consent

SUMMARY:
SUMMARY:

The purpose of this study is to learn how to better educate patients about oral health procedures and treatments through an improved informed consent process. We will gather information from patients and health care providers, and design and test a computerized consent system called SmartConsent.

HYPOTHESIS:

1. Subjects who use SmartConsent will have increased knowledge (cognitive achievement) about oral health disease and treatment than patients who view the standard consent
2. Subjects who use SmartConsent will have less decisional conflict in their decision regarding an oral health procedure than those who view the standard consent form
3. Subjects who use SmartConsent will have greater visit satisfactions scores than those who view the standard consent form

DETAILED DESCRIPTION:
Communicating personalized information to patients about the risks, benefits and other critical information about dental disease and treatment is often difficult for providers. In this proposal we seek to develop a novel informed consent system that can accurately translate and communicate information to patients in a standardized and effective manner based on their diagnosis and prescribed treatment. We aim to integrate SmartConsent into the institutional electronic patient record (EPR). This research is translational as it seeks to determine how providers can better communicate information to patients so they can make appropriate decisions about dental treatments and options.

The advent of electronic health records allows an informed consent document to be automatically personalized based on a patient's demographic profile, literacy level, language preference, and prior medical history. A computerized consent also allows the presentation of information in a format beyond text such as through the use of multimedia. Further, in a computer-based consent, we can quickly test a patient's knowledge about a diagnosis and procedure to ensure that key information has been delivered. In this proposal we seek to discover if a computer-based informed consent is more effective in educating patients about common oral health disease and treatment (e.g., reason for extracting a tooth, causes of periodontal disease, risks associated with dental implants). We also seek to determine its feasibility in a real clinical practice by measuring time taken and impact on workflow compared to the traditional consent process.

ELIGIBILITY:
Inclusion Criteria:

* Adult
* English-speaking
* Diagnosis of pulpal disease

Exclusion Criteria:

* Treatment required referral outside of clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Urgent Care Clinic at UT Dental Branch at Houston
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2013-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Valenza, DDS, Principal Investigator — UTHSC-Houston